CLINICAL TRIAL: NCT03110627
Title: Increasing Detection of Sub-Clinical Atrial Fibrillation in Defibrillator Patients With the Use of a VDD-ICD Lead: The Dx-AF Study
Brief Title: Increasing Detection of Sub-Clinical Atrial Fibrillation in Defibrillator Patients With the Use of a VDD-ICD Lead
Acronym: Dx-AF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Unity Health Toronto (Other)
Collaborators: Applied Health Research Centre (Other); Biotronik Canada Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: Dx01
Record Dates: First submitted 2017-04-07; First posted 2017-04-12 (Actual); Last update posted 2021-04-30 (Actual); Status verified 2021-04

CONDITIONS: Cardiac Arrhythmias; Atrial Fibrillation and Flutter; Cardiovascular Diseases; Implantable Cardioverter-Defibrillators
Keywords: Single-chamber ICD (implantable cardioverter-defibrillator); Cardiac Arrhythmias; Atrial fibrillation; Atrial flutter; Stroke
MeSH Terms: conditions — Arrhythmias, Cardiac; Atrial Fibrillation; Cardiovascular Diseases; Atrial Flutter; Stroke | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: DX AF is a prospective, randomized-controlled, open-label trial. Patients who are identified on clinical grounds for a single-chamber ICD will randomized to a VDD ICD (experimental group) or single chamber ICD (control group).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VDD ICD (Experimental): VDD ICD - A single-lead ICD system with the ability to sense atrial rhythm from the floating electrode (a VDD-ICD known as the DX) - Experimental group
  Interventions: Device: VDD ICD (experimental group)
- VVI ICD (Active Comparator): VVI ICD - Single chamber ICD system - Control group
  Interventions: Device: Single chamber VVI ICD (control group)

INTERVENTIONS:
Device: VDD ICD (experimental group) — Patients who are identified on clinical grounds for a single-chamber ICD will randomized to a VDD ICD (experimental group) or single chamber ICD (control group).
  The study will compare the Dx-ICD system (experimental) to standard VVI-ICD (control) on the ability to diagnose silent AF in patients without prior AF receiving an ICD for standard indications.
  Other Names: Experimental: DX ICD (experimental group)
  Arms: VDD ICD
Device: Single chamber VVI ICD (control group) — Patients who are identified on clinical grounds for a single-chamber ICD will randomized to a VDD ICD (experimental group) or single chamber ICD (control group).
  The study will compare the Dx-ICD system (experimental) to standard VVI-ICD (control) on the ability to diagnose silent AF in patients without prior AF receiving an ICD for standard indications.
  Other Names: Control: Single chamber VVI ICD
  Arms: VVI ICD

SUMMARY:
This study aims to compare the Dx-ICD system (experimental) to standard VVI-ICD (control) on the ability to diagnose silent AF in patients without prior AF receiving an ICD for standard indications.

DETAILED DESCRIPTION:
Recipients of implantable defibrillators (ICD) are at high risk of developing both AF and stroke, given the presence of multiple cardiovascular risk factors. Oral anticoagulation can prevent most strokes in patients with AF; provided that AF is recognized before a stroke occurs. Up to about 40% of incident AF may be sub-clinical, producing minimal or no symptoms, or being too short to allow detection.

DX AF is a prospective, randomized-controlled, open-label trial. Patients who are identified on clinical grounds for a single-chamber ICD will be randomized to a VDD ICD (experimental group) or single chamber ICD (control group).

The study will compare the Dx-ICD system (experimental) to standard VVI-ICD (control) on the ability to diagnose silent AF in patients without prior AF receiving an ICD for standard indications.

ELIGIBILITY:
Inclusion Criteria:

* Patients with ischemic or non-ischemic cardiomyopathy,
* LVEF<50%, scheduled for primary or secondary prevention ICD
* Treating physicians feel that the use of single chamber ICD is appropriate
* No ECG-documented history of AF or flutter
* Age > 50 years

Exclusion Criteria:

* Known AF or flutter
* Current use of class I or III anti-arrhythmic medications
* Participants unwilling to attend study follow-up visits, considered unreliable for compliance or with an anticipated life expectancy less than 3 years

Min Age: 51 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 188 (Actual)
Dates: Start 2017-03-31 (Actual); Primary Completion 2022-03-31 (Estimated); Study Completion 2022-03-31 (Estimated)

PRIMARY OUTCOMES:
Atrial Fibrillation or atrial flutter lasting at least 6 minutes | During the entire time of follow up - 3 years
  Atrial Fibrillation or atrial flutter lasting at least 6 minutes detected by the ICD, ECG, Holter monitor or telemetry.

SECONDARY OUTCOMES:
Need for any ICD lead repositioning or replacement | 60 days
  Composite outcome of serious device-related complications occurring in the 60 days from the time of ICD insertion.
Pneumothorax | 60 days
  Composite outcome of serious device-related complications occurring in the 60 days from the time of ICD insertion.
New pericardial effusion | 60 days
  Composite outcome of serious device-related complications occurring in the 60 days from the time of ICD insertion.
Cardiac tamponade | 60 days
  Composite outcome of serious device-related complications occurring in the 60 days from the time of ICD insertion.
Procedure-related death or wound infection | 60 days
  Composite outcome of serious device-related complications occurring in the 60 days from the time of ICD insertion.

CONTACTS AND LOCATIONS:
Overall Officials: Eugene Crystal, MD, FRCP(C), Principal Investigator — Sunnybrook Health Sciences Centre
Locations (9):
- Canada (9):
  - Royal Alexandra Hospital, Edmonton, Alberta
  - Vancouver Island Health Authority, Vancouver, British Columbia
  - Saint John Regional Hospital, Saint John, New Brunswick
  - Health Sciences North, Greater Sudbury, Ontario
  - Scarborough and Rouge Hospital - Centenary Site, Toronto, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - IUCPQ - Institut universitaire de cardiologie et de pneumologie de Québec, Laval, Quebec
  - HSCM - L'Hôpital du Sacré-Coeur de Montréal, Montreal, Quebec
  - CHUS - Centre Hospitalier Universitaire de Sherbrooke, Sherbrooke, Quebec

IPD SHARING:
Plan to Share IPD: No